CLINICAL TRIAL: NCT01043120
Title: A Randomised, Double-blind, Parallel Groups, Placebo-controlled, Multi-centre Trial in Oocyte Donors Assessing the Effects of Barusiban, a Selective Oxytocin Antagonist, on Uterine Contractions on the Day of Embryo Transfer
Brief Title: Effect of Oxytocin Antagonist on Reduction of Uterine Contractions
Acronym: EFFORT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FE200440 CS11; 2009-012323-29
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: In Vitro Fertilisation (IVF) Treatment
MeSH Terms: interventions — barusiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Barusiban (Experimental)
  Interventions: Drug: Barusiban
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Barusiban — IV bolus of 20 mg for 1 minute followed by an IV infusion of 19 mg for up to 59 minutes. The maximum total duration of administration was 60 minutes.
  Arms: Barusiban
Drug: Placebo — IV bolus of saline (sodium chloride 0.9%) for 1 minute followed by an IV infusion of saline (sodium chloride 0.9%) for up to 59 minutes. Details on injection volume, infusion rates and doses are tabulated below.
  Arms: Placebo

SUMMARY:
The main purpose of this clinical research trial was to evaluate the effects of barusiban compared to placebo on uterine contractions on luteal phase uterine contractions in oocyte donors supplemented with progesterone.

DETAILED DESCRIPTION:
This was a randomised, double-blind, parallel groups, placebo-controlled, multi-centre trial. It was designed to evaluate the efficacy of barusiban, a selective oxytocin antagonist, on reducing the frequency of uterine contractions on the day of embryo transfer.

Participants in this trial were oocyte donors who had undergone controlled ovarian hyperstimulation in the long gonadotrophin-releasing hormone (GnRH) agonist protocol or the multiple-dose GnRH antagonist protocol, had received human chorionic gonadotrophin (hCG) for triggering of final follicular maturation and had undergone oocyte retrieval (OR) with a yield of ≥ 6 cumulus-oocyte-complexes. The duration of the trial was two days: Day OR +2 (screening, randomisation and dosing of investigational medicinal product) and Day OR +3 (end-of-trial).

On Day OR +2, participants were screened and subsequently randomised to barusiban or placebo. All participants received an intravenous (IV) bolus for 1 minute followed by an IV infusion for up to 59 minutes, administered via an indwelling catheter, of barusiban or placebo. Bolus volume and infusion rate were identical for barusiban and placebo. A mock embryo transfer (MET) procedure was performed 40 minutes after start of dosing and included intrauterine administration of a non-radioactive ultrasound contrast agent (SONOVUE) via the embryo transfer catheter. Transvaginal ultrasound of around 5 minutes duration was performed at seven time points on Day OR +2 and covered a span of approximately 2.5 hours including pre-dosing, during dosing, before and after mock embryo transfer, and post-dosing. The transvaginal ultrasound recordings were analysed for frequency of uterine contractions and other uterine contractility parameters by a central independent assessor, blinded to treatment allocation. Movement of the ultrasound contrast agent after the mock embryo transfer procedure was evaluated by the central independent assessor.

As an attempt to document the impact of uterine contractions on potential embryo expulsion, an exploratory evaluation of the movement of an ultrasound contrast agent (SONOVUE)administered intrauterinely via an embryo transfer catheter during the mock embryo transfer was performed. The anatomical point of release of the ultrasound contrast agent (correct or incorrect deposition site, and estimated distance from fundus) as well as any immediate movement (yes/no) of the bolus was recorded by the central independent assessor.

Definitions:

The frequency of uterine contractions was defined as the number of uterine contractions per minute. A contraction was defined as one sequential upward and downward vertical displacement of the endometrial / myometrial interface over time. The frequency was the inverse of period converted to contractions per minute.

The period was the average time it took to complete one contraction during the studied time interval. It was calculated from both the peaks and the troughs at the anterior and posterior endometrial /myometrial interfaces. The period was measured in seconds per contraction.

The external contractile measure was the mean wave amplitude in mm at the lumenal surface. This metric was measured at the lumenal peaks and troughs only and was a measurement designed to study the relationship between endometrial wave activity, manifest as bulk motion of the uterus, versus internal contractile strength. The external contractile measure was reported in mm/contraction. The external contractile measure quantified the movement of the uterus as a whole as measured at the lumen, i.e. the motion of the uterus relative to the body.

The internal contractile measure was the strength of the contractions based upon the sum of the contraction amplitudes measured at the anterior and posterior endometrial / myometrial interfaces. The amplitude at each interface was defined as the average difference between the endometrial / myometrial-lumenal distance measured at the peaks and troughs of the endometrial / myometrial interfaces. The internal contractile measure was reported in mm/contraction. The internal contractile measure quantified the movement of the endometrium relative to the lumen, i.e. the motion internal to the uterus.

The total contractile measure was the sum of the external contractile measure and the internal contractile measure and quantified total muscle movement in the uterus. If the waves at the anterior and posterior endometrial / myometrial interfaces were in phase then there was no endometrial motion relative to the lumen and the motion was a pure wave motion with the internal contractile measure equal to zero. The total contractile measure was reported in mm/contraction.

Inter-subendometrial space was measured clinically as the distance between the anterior stratum basalis and posterior stratum basalis layers in mid-sagittal plane at an anatomic location between 5 and 10 mm from the fundus. All clinical inter-subendometrial space measurements were made by selecting a clear image of the uterus, waiting for any contractions to pass and freezing the image.

A linear distance measurement was then taken between the anatomic landmarks described above. Inter-subendometrial space was calculated from existing measurements using the mean of all measurements identifying the endometrial-myometrial interfaces on the superior and inferior surfaces in each endometrial strip when the arrows identifying endometrial contractions were placed for motion analysis. Inter-subendometrial space was reported in mm.

The direction of wave propagation was classified as one of the following:

* Fundal (from cervix to fundus)
* Cervical (from fundus to cervix)
* Convergent (opposing) starting simultaneously from cervix and fundus
* Focal local contractions (which are not involving the whole uterine walls)
* No activity
* NE: not evaluable At each assessment time point, the most predominant type of direction of wave propagation was recorded.

Dispersion of the ultrasound contrast agent bolus after release from the catheter was recorded as yes/no and number of dispersed fragments, if applicable.

Location of the ultrasound contrast agent bolus was categorised as follows:

* Upper 1/3 (fundal) part of uterine cavity
* Central 1/3 of uterine cavity
* Lower 1/3 (cervical) part of the uterine cavity
* Intralumenal part of Fallopian tube
* Intra-cervical
* Vaginal
* NE: not evaluable Distance from the apex of the fundus at the myometrial-endometrial interface to the position of the microdroplet of ultrasound contrast agent was recorded in mm.

Velocity of the bolus of ultrasound contrast agent was assessed from distance and time, and was recorded in mm/hour.

ELIGIBILITY:
Participants eligible for this trial were oocyte donors 18-37 years of age, who had undergone controlled ovarian hyperstimulation in the long GnRH agonist protocol or the multiple-dose or single-dose GnRH antagonist protocols, had received hCG (10,000 IU urinary hCG or 250 μg recombinant hCG) for triggering of final follicular maturation and had undergone oocyte retrieval. Participants had given signed informed consent, were generally healthy and with a body mass index (BMI) of 18.5-29 kg/m2.

Participants were excluded in case of endometriosis stage I-IV or uterine pathology. Participants were willing to not have intake of alcoholic beverages during the trial, to not have sexual intercourse during the trial, and to either maintain sexual abstinence or use a highly effective method of contraception from end-of-trial till onset of next menses.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Frequency of uterine contractions, Intention-To-Treat (ITT) Analysis Set | 30 minutes after start of dosing
  Frequency of uterine contractions was assessed by transvaginal ultrasound. The transvaginal ultrasound recordings were analysed for uterine contractions by a central independent assessor, blinded to treatment allocation.
Frequency of uterine contractions, Per-Protocol (PP) Analysis Set | 30 minutes after start of dosing
  Frequency of uterine contractions was assessed by transvaginal ultrasound. The transvaginal ultrasound recordings were analysed for uterine contractions by a central independent assessor, blinded to treatment allocation.

SECONDARY OUTCOMES:
Uterine contractile measures | During and after dosing (one day)
Inter-endometrial space | 30 minutes after start of dosing
Direction of Wave Propagation
Direction of Wave Propagation, Post-hoc analysis | 30 min after start of dosing and MET
  Post-hoc analyses of the secondary endpoint parameter wave propagation were conducted. The ability of the contractile waves to propagate uterine contractions after mock embryo transfer was categorised (No, Yes, Indeterminate, NA or NE) by the central assessor for the following time points: Pre-dose, 30 min after start of dosing and at end of mock embryo transfer (MET0 min). Fisher's exact p-value test comparing the distribution of No and Yes between treatment groups was performed
Dispersion, Location, Distance from Point of Release and Velocity of Ultrasound Contrast Agent

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (5):
- UZ Brussel, Brussels, Belgium
- Czechia (2):
  - IVF Institute, Pilsen
  - ISCARE IVF a.s., Prague
- Spain (2):
  - IU Dexeus, Barcelona
  - IVI Madrid, Madrid